CLINICAL TRIAL: NCT00004916
Title: Phase I/II Study of Mesna, Ifosfamide, Teniposide and Weekly Taxol (MITTen) in Relapsed Lymphoma
Brief Title: Ifosfamide, Teniposide, and Paclitaxel in Treating Patients With Relapsed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 98H2; NU-98H2; NCI-G00-1711
Record Dates: First submitted 2000-03-07; First posted 2003-05-14 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma | interventions — Ifosfamide; Paclitaxel; Teniposide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ifosfamide
Drug: paclitaxel
Drug: teniposide
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of ifosfamide, teniposide, and paclitaxel in treating patients who have relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicities associated with the combination of ifosfamide, teniposide, and weekly paclitaxel in patients with relapsed non-Hodgkin's lymphoma.
* Evaluate response rate and time to disease progression in these patients treated with this regimen.

OUTLINE: This is a dose escalation study of teniposide. Patients are stratified according to whether they proceed to stem cell transplant or not.

Patients receive ifosfamide IV over 1-2 hours on days 1-3 every 3 weeks, teniposide IV over 2 hours on day 1 every 3 weeks, and paclitaxel IV over 1 hour weekly. Patients who are not candidates for stem cell transplant continue treatment for 120 days in the absence of disease progression or unacceptable toxicity. Patients proceeding to stem cell transplant continue treatment for 36 days. Peripheral blood stem cells (PBSC) may be harvested at this time if autologous transplant is planned. Transplant patients may then continue with chemotherapy or proceed to autologous or allogeneic PBSC transplant.

Cohorts of 3-5 patients receive escalating doses of teniposide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 5 patients experience dose limiting toxicities.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 15-50 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intermediate or high grade non-Hodgkin's lymphoma

  * No lymphoblastic or small cleaved lymphoma
* Progressive disease following doxorubicin based chemotherapy

  * No more than 2 prior treatment regimens
* Measurable or evaluable disease NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No significant cardiac disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active or uncontrolled second malignancy
* No other medical problems that would preclude therapy
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior stem cell transplant allowed

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo I. Gordon, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States